CLINICAL TRIAL: NCT01308749
Title: A Pilot Study of Oxytocin in Children and Adolescents With Autistic Disorder
Brief Title: A Study of Oxytocin in Children and Adolescents With Autistic Disorder
Acronym: Oxytocin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-0493
Record Dates: First submitted 2011-02-28; First posted 2011-03-04 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Intervention: Drug: placebo
  Interventions: Drug: Placebo
- Oxytocin (Active Comparator): Intervention: Drug: Syntocinon® Nasal Spray
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Subjects will use the Syntocinon® Nasal Spray (oxytocin) twice daily for 8 weeks if they are randomized to that arm in the Randomized Phase. All subjects will use the Syntocinon® Nasal Spray twice daily for 8 weeks in the Open Label Phase.
  Subjects ages 3-10 years old will be titrated up to a maximum dose of 24 International units (IU). Subjects ages 11-17 years old will be titrated up to a maximum dose of 32IU.
  Other Names: Syntocinon® Nasal Spray
  Arms: Oxytocin
Drug: Placebo — Placebo Nasal Spray
  Arms: Placebo

SUMMARY:
The investigators propose to conduct this pilot study to evaluate oxytocin as a supplemental treatment for improving social difficulties in individuals with autism.

DETAILED DESCRIPTION:
The proposed pilot study is an essential first step toward rigorously evaluating oxytocin treatment of individuals with autism. The biologic actions of oxytocin on social cognition and prosocial behaviors and the clinical, genetic and epigenetic evidence for involvement of the oxytocin system in the pathophysiology of some cases of autism strongly suggest that supplemental oxytocin therapy could significantly improve the social disabilities involved in autism. Many people feel that these social difficulties are the most characteristic and central feature of autism. Overall, this study aims to determine the tolerability, accessibility, and feasibility of an oxytocin pilot study.

This study will consent up to 30 subjects in order to randomize up to 25 subjects into a 2-month (8 weeks) randomized double-blind, placebo-controlled initial treatment period, a subsequent 2-month (8 weeks) period in which all participants receive oxytocin, and up to three post-treatment visits that occur at week 28 (±2 weeks),an interim visit anytime between week 16 and week 76 only for those patients who plan to start oxytocin on their own outside of study treatment and who will experience a lag time between week 16 (end of open label treatment) and when outside oxytocin treatment will begin, and some time before week 76. The investigators hope that this study will help to inform future study designs in determining whether a short term or long term treatment trial is necessary to observe significant effects. This will also help to develop systematic preliminary safety measures.

ELIGIBILITY:
Inclusion Criteria:

* Between 3 and 17 years old, inclusive.
* Have a clinical diagnosis of autistic disorder confirmed according to Diagnostic Statistical Manual of Mental Disorders-IV criteria by using the Autism Diagnostic Interview - Revised (ADI-R) and/or the Autism Diagnostic Observation Scale (ADOS, Lord et al., 1989).

Exclusion Criteria:

* Changes in allied health therapies, behavioral or educational interventions within the past 2 months of the baseline visit other than those associated with school holidays.
* Changes in psychotropic and alternative medication doses in the last 30 days of the baseline visit.
* Subjects with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. This includes, but is not limited to, Rett Syndrome, impairment of renal function, evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder and uncontrolled hypertension), respiratory, hepatic, or gastrointestinal disease.
* Marked sensory impairment such as deafness or blindness that would interfere with conduct of the study.
* Pregnancy/Nursing because of the unknown effects of oxytocin to unborn babies and/or nursing infants. All females of child-bearing potential will be administered a urine or serum pregnancy test at screening and at any point during the study at physician discretion. Refusal to undergo a pregnancy test will result in exclusion from the study. The investigators will share results of pregnancy test with the subject's legal guardian.
* Refusal to practice contraception if sexually active because the effects of exposure to high concentrations of oxytocin on sperm or newly conceived embryos are unknown. Sexually active men and women should not take part in this study if they and their partners are not both using an effective birth control method (for example, women use birth control pills, an intrauterine device (IUD) or a diaphragm and men use condoms).
* Inability of caretakers to speak English.
* Absence of a consistent caretaker to report on symptoms.
* Subjects who, in the Investigator's opinion, might not be suitable for the study.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a 2 sequence (arm) study with 2 periods - double-blind (0-8 weeks) and open label (8-16 weeks). The sequences are 1: oxytocin-oxytocin and 2: placebo-oxytocin. 1 participant from sequence 1 did not enter period 2 due to withdrawal due to adverse events.
Groups:
- Sequence 1: Oxytocin-oxytocin: 8 weeks of double blind oxytocin followed by 8 weeks of open label oxytocin
- jSequence 2: Placebo-oxytocin: 8 weeks of of double blind placebo followed by 8 weeks of open-label oxytocin; this is the control group
Period: Period 1: Double Blind Treatment
Arm/Group | Sequence 1: Oxytocin-oxytocin | jSequence 2: Placebo-oxytocin
Started | 12 | 13
Completed | 11 | 13
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2: Open Label Treatment
Arm/Group | Sequence 1: Oxytocin-oxytocin | jSequence 2: Placebo-oxytocin
Started | 11 | 13
Completed | 11 | 11
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The one participant in the oxytocin group who dropped out after 2 days is not included in the demographics or outcome analyses since no post baseline data other than AEs was obtained. This participant is included in the AE analysis.
Groups:
- Sequence 2:Placebo-oxytocin: Intervention: Drug: placebo
  Placebo: Placebo Nasal Spray
- Sequence 1: Oxytocin-oxytocin: Intervention: Drug: Syntocinon® Nasal Spray
  Oxytocin: Subjects will use the Syntocinon® Nasal Spray (oxytocin) twice daily for 8 weeks if they are randomized to that arm in the Randomized Phase. All subjects will use the Syntocinon® Nasal Spray twice daily for 8 weeks in the Open Label Phase.
  Subjects ages 3-10 years old will be titrated up to a maximum dose of 24 international units (IU). Subjects ages 11-17 years old will be titrated up to a maximum dose of 32IU.
- Total: Total of all reporting groups
Arm/Group | Sequence 2:Placebo-oxytocin | Sequence 1: Oxytocin-oxytocin | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 12 | 25
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (4.4) | 10.6 (4.4) | 10.3 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Non-verbal [Count of Participants; unit: Participants] | 7 | 4 | 11
Intelligence Quotient (IQ) <70 [Count of Participants; unit: Participants] | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Could Tolerate Twice Daily Oxytocin
Description: This study will help to determine tolerability of intranasal oxytocin treatment in children with autism by measuring the ability of at least 80% of the sample to tolerate twice daily intranasal administration of oxytocin.
Time Frame: Week 0 to week 8
Population: This is over period 1, the double blind phase (week 0 to week 8) only
Measure: Count of Participants; unit: Participants
Groups:
- Sequence 2: Placebo:Oxytocin: Intervention: Drug: placebo double blind for 8 weeks then oxytocin open label for 8 weeks
- Sequence 1: Oxytocin:Oxytocin: Intervention: Drug: oxytocin = Syntocinon® Nasal Spray
  total of 16 weeks exposure Subjects ages 3-10 years old will be titrated up to a maximum dose of 24IU. Subjects ages 11-17 years old will be titrated up to a maximum dose of 32IU.
Arm/Group | Sequence 2: Placebo:Oxytocin | Sequence 1: Oxytocin:Oxytocin
Number analyzed (Participants) | 13 | 12
Participants | 13 | 11
Statistical Analysis 1: Comparison: Sequence 2: Placebo:Oxytocin vs Sequence 1: Oxytocin:Oxytocin; Test type: Other; No analyses were completed, this is descriptive only and is an absolute value (number of participants)

2. Primary Outcome: Number of Participants Who Could Tolerate Twice Daily Oxytocin
Description: as for outcome 1
Time Frame: Week 0 to week 16
Population: all participants who recieved oxytocin at any time
Measure: Count of Participants; unit: Participants
Groups:
- Sequence 2: Placebo:Oxytocin: This is accounts for participants from week 0 to week 16. All participants first received placebo (week 0 to week 8) and then subsequently received oxytocin (week 8 to week 16)
- Sequence 2: Oxytocin:Oxytocin: This accounts for all participants starting from baseline to week 16 who received oxytocin the whole time. All participants participants received oxytocin for the full 16 weeks.
Arm/Group | Sequence 2: Placebo:Oxytocin | Sequence 2: Oxytocin:Oxytocin
Number analyzed (Participants) | 13 | 12
Participants | 11 | 11

3. Secondary Outcome: Change in Mean Plasma Oxytocin Level During Period 1 - Double Blind Phase
Description: Blood samples will be collected to obtain proof of concept data regarding changes in afternoon plasma oxytocin levels
Time Frame: Week 0 to week 8
Population: participants with oxytocin plasma levels at baseline and week 8
Measure: Mean (Standard Deviation); unit: picograms/mL (pg/mL)
Groups:
- Sequence 2: Placebo:Oxytocin: sequence2: placebo:oxytocin
  Placebo: Placebo Nasal Spray
- Sequence 1: Oxytocin:Oxytocin: Intervention: Drug: Syntocinon® Nasal Spray
  Oxytocin: Subjects will use the Syntocinon® Nasal Spray (oxytocin) twice daily for 8 weeks if they are randomized to that arm in the Randomized Phase. All subjects will use the Syntocinon® Nasal Spray twice daily for 8 weeks in the Open Label Phase.
  Subjects ages 3-10 years old will be titrated up to a maximum dose of 24IU. Subjects ages 11-17 years old will be titrated up to a maximum dose of 32IU.
Arm/Group | Sequence 2: Placebo:Oxytocin | Sequence 1: Oxytocin:Oxytocin
Number analyzed (Participants) | 11 | 10
picograms/mL (pg/mL) | -0.69 (1.69) | -0.15 (1.53)

4. Secondary Outcome: Change in Mean Weight
Description: changes during period 1
Time Frame: between weeks 0 and 8
Population: The subject who discontinued after 2 days did not have repeat assessments and is excluded from these analyses
Measure: Mean (Standard Error); unit: pounds
Groups:
- Sequence 1: Oxytocin-oxytocin: Intervention: Drug: Syntocinon® Nasal Spray
  Oxytocin: Subjects will use the Syntocinon® Nasal Spray (oxytocin) twice daily for 8 weeks if they are randomized to that arm in the Randomized Phase. All subjects will use the Syntocinon® Nasal Spray twice daily for 8 weeks in the Open Label Phase.
  Subjects ages 3-10 years old will be titrated up to a maximum dose of 24IU. Subjects ages 11-17 years old will be titrated up to a maximum dose of 32IU.
- Sequence 2: Placebo :Oxytocin: Intervention: Drug: placebo
  Placebo: Placebo Nasal Spray
Arm/Group | Sequence 1: Oxytocin-oxytocin | Sequence 2: Placebo :Oxytocin
Number analyzed (Participants) | 11 | 13
pounds | 1.4 (1.3) | 2.4 (0.7)

5. Secondary Outcome: Change in Mean Total Social Social Responsiveness Scale (SRS) T-score
Description: The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The raw score of each individual item is summed to create a total raw score. The total raw score is then translated into a total T-scores (which are the equivalent of standard scores). Total T-scores results are as follows: 59 and below: within normal limits, 60-65: Mild range of impairment 66-75: Moderate range of impairment 76 or higher: Severe range of impairment.
Time Frame: 0-8 weeks, blinded treatment, period 1
Population: All participants with at least one post baseline assessment, 1 person from sequence 1 discontinued due to no post baseline measures
Measure: Mean (Standard Error); unit: T-scores
Groups:
- Sequence 2: Placebo :Oxytocin: placebo x8 weeks then oxytocin x 8weeks
Arm/Group | Sequence 1: Oxytocin-oxytocin | Sequence 2: Placebo :Oxytocin
Number analyzed (Participants) | 11 | 13
T-scores | -5.1 (2.3) | -3.9 (3.3)
Statistical Analysis 1: Comparison: Sequence 1: Oxytocin-oxytocin vs Sequence 2: Placebo :Oxytocin; Test type: Equivalence — Within group test of difference using t-scores adjusted by baseline score, no correction for multiple comparisons, nonparametric model; p = 0.023, t-test, 2 sided

6. Secondary Outcome: Change in Mean Autism Diagnostic Observation Schedule (ADOS) Total Score
Description: The ADOS is a semi-structured assessment used to assess and diagnose individuals suspected of having autism of varying ages, developmental levels, and language skills (from no speech to verbally fluent). The ADOS includes four modules, each requiring just 35-40 minutes to administer. The individual being evaluated is given just one of 4 modules, depending on his or her expressive language level and chronological age. The rater will observe social and communication behaviors during various activities in the appropriate module. A rater then uses a 0-3 scale to rate each type of behavior. A select number of individual items will be summed for a total score representing communication and reciprocal social interaction. In scoring all 3's are collapsed to a 2. A higher score indicates more severe impairment. Ranges of scores are as follows: Module 1: 0-24, Module 2: 0-24, Module 3: 0-22, Module 4: 0-22.
Time Frame: Baseline to 16 Weeks
Population: 1 patient without post baseline measures is not included
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Sequence 1: Oxytocin-oxytocin | Sequence 2: Placebo :Oxytocin
Number analyzed (Participants) | 11 | 13
scores on a scale | -0.36 (0.39) | -0.31 (0.29)

7. Secondary Outcome: Change in Mean Aberrant Behavior Checklist (ABC)-Social Withdrawal Subscale Score Over Both Periods
Description: Efficacy measures included the Aberrant Behavior Checklist -Social Withdrawal subscale scor. The ABC which focuses on problem behaviors in five subdomains, including irritability, attention, repetitive behaviors, unusual speech, and lethargy. A modified version of the lethargy subscale was used. Typically the Lethargy subscale includes 16 items, however, for our purposes 3 items that were specifically related to lethargy (i.e.: listlessness) were removed so that the focus could primarily be on aberrant social behavior. Differences in only the Social Withdrawal domain were assessed.The is the sum of items, each rated among 0 = Not at all; 1 = Slight in degree; 2 = Moderately serious; and 3 = Severe in degree. The ABC- Social Withdrawal total score ranges from 0 to 39. Higher values represent greater severity of illness.
Time Frame: Baseline to 16 Weeks
Population: population of participants with all data available for mixed models analysis no data carried forward
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Sequence 1: Oxytocin-oxytocin | Sequence 2: Placebo :Oxytocin
Number analyzed (Participants) | 11 | 11
scores on a scale | -3.7 (1.0) | -2.2 (1.9)
Statistical Analysis 1: Comparison: Sequence 1: Oxytocin-oxytocin vs Sequence 2: Placebo :Oxytocin; Test type: Equivalence — t-test between groups; p = 0.23, t-test, 2 sided; no adjustment for multiple comparison. non parametric

8. Secondary Outcome: Change in Mean Pervasive Developmental Disorder Behavior Inventory - Screening Version (PDDBI-SV) Total Score Over Both Periods
Description: The PDDBI-SV examines both adaptive and maladaptive behaviors related to autism. It has normative scores for children between 2-11 years. For children 12 years and older, the norms (11 years, 11 months) will be used. Each item is scored on a scale from 0-3. For the first 9 items, the total of individual items is summed. For items 10-18, the scores are reversed and then summed (i.e.: 0=3, 1 =2, 2=2, 3 = 0). Then the total of 0-9 and then the reversed scored items 10-18 are summed for a final total score. Higher scores indicate more impairment. The range of total scores is 0-54. ASD/Social deficits unlikely: 0-6, More information needed/borderline: 7-10, autism spectrum disorder (ASD)/social deficits likely (mild):11-14, ASD/social deficits likely (moderate): 15-29, ASD/social deficits likely (severe): 30-37, ASD/social deficits likely (extreme): 38 or higher.
Time Frame: Baseline to 16 Weeks
Population: used only subjects with all data points no data carried forward
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Sequence 1: Oxytocin-oxytocin | Sequence 2: Placebo :Oxytocin
Number analyzed (Participants) | 11 | 11
scores on a scale | -3.6 (2.4) | -3.0 (2.2)

9. Secondary Outcome: Change in Mean Systolic Blood Pressure During Period 1
Description: Change in mean systolic blood pressure during double blind phase
Time Frame: Week 0 to 8
Population: The one subject who discontinued at week 1 did not have follow up data to include in the analysis.
Measure: Mean (Standard Error); unit: millimeters of mercury (mmHg)
Groups:
- Sequence 1: Oxytocin-oxytocin: 8 weeks of Intervention: Drug: oxytocin (Syntocinon) baseline to week 8
- Sequence 2: Placebo :Oxytocin: Subjects who received 8 weeks of placebo treatment (baseline to week 8)
Arm/Group | Sequence 1: Oxytocin-oxytocin | Sequence 2: Placebo :Oxytocin
Number analyzed (Participants) | 11 | 13
millimeters of mercury (mmHg) | -7.6 (2.8) | 1.5 (3.2)

10. Secondary Outcome: Mean Change in Prolactin Levels Over Period 1
Description: Serum prolactin levels were collected and analyzed in participants
Time Frame: Week 0 to 8
Measure: Mean (Standard Error); unit: nanograms per milliliter (ng/mL)
Groups:
- Sequence 1: Oxytocin-oxytocin: 8 weeks of Intervention following randomization
- Sequence 2: Placebo :Oxytocin: 8 weeks double blind placebo followed by 8 wks open label oxytocin
Arm/Group | Sequence 1: Oxytocin-oxytocin | Sequence 2: Placebo :Oxytocin
Number analyzed (Participants) | 11 | 13
nanograms per milliliter (ng/mL) | -3.6 (2.68) | 1.17 (1.63)

11. Secondary Outcome: Mean Change in Temperature During Period 1
Description: Temperature was collected on each participant via oral or temporal thermometer. The mean change in each group was assessed.
Time Frame: Week 0 to 8
Measure: Mean (Standard Error); unit: degrees fahrenheit
Groups:
- Sequence 2: Placebo :Oxytocin: 8 weeks of intervention following randomization
Arm/Group | Sequence 1: Oxytocin-oxytocin | Sequence 2: Placebo :Oxytocin
Number analyzed (Participants) | 11 | 13
degrees fahrenheit | -0.7 (0.2) | -0.1 (0.2)

ADVERSE EVENTS:
Time Frame: Period 1 0-8 weeks comparing sequence 1 and 2, Period 2 comparing sequence1 and 2
Groups:
- Sequence 1: Oxytocin:Oxytocin Period 1weeks 0-8: Intervention: Drug: Syntocinon® Nasal Spray
  Oxytocin: Subjects will use the Syntocinon® Nasal Spray (oxytocin) twice daily for 8 weeks if they are randomized to that arm in the Randomized Phase. All subjects will use the Syntocinon® Nasal Spray twice daily for 8 weeks in the Open Label Phase.
  Subjects ages 3-10 years old will be titrated up to a maximum dose of 24IU. Subjects ages 11-17 years old will be titrated up to a maximum dose of 32IU.
- Sequence 2: Placebo: Oxytocin Period 1 Weeks 0-8: Intervention: Drug: placebo
  Placebo: Placebo Nasal Spray
- Sequence 1: Oxytocin:Oxytocin Period 2, Weeks 8-16: evaluates longer term adverse events with oxytocin
- Sequence 2: Placebo:Oxytocin Period 2: evaluates acute exposure to oxytocin in sequence 2 participants
Arm/Group | Sequence 1: Oxytocin:Oxytocin Period 1weeks 0-8 | Sequence 2: Placebo: Oxytocin Period 1 Weeks 0-8 | Sequence 1: Oxytocin:Oxytocin Period 2, Weeks 8-16 | Sequence 2: Placebo:Oxytocin Period 2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/13 | 0/24 | 0/13
Other Adverse Events (participants affected / at risk) | 12/12 | 10/13 | 8/11 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sequence 1: Oxytocin:Oxytocin Period 1weeks 0-8 (N=12) | Sequence 2: Placebo: Oxytocin Period 1 Weeks 0-8 (N=13) | Sequence 1: Oxytocin:Oxytocin Period 2, Weeks 8-16 (N=24) | Sequence 2: Placebo:Oxytocin Period 2 (N=13)
Croup (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0/11 (0) | 0 (0) — unanticipated, unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1: Oxytocin:Oxytocin Period 1weeks 0-8 (N=12) | Sequence 2: Placebo: Oxytocin Period 1 Weeks 0-8 (N=13) | Sequence 1: Oxytocin:Oxytocin Period 2, Weeks 8-16 (N=11) | Sequence 2: Placebo:Oxytocin Period 2 (N=13)
# of participants with any adverse event (General disorders) | 12 (59) | 10 (53) | 7 (19) | 12 (46)
# with moderate adverse event (General disorders) | 5 (16) | 9 (20) | 3 (5) | 6 (16)
# with severe adverse event (General disorders) | 5 (12) | 2 (6) | 1 (3) | 1 (5)
insomnia (Nervous system disorders) | 4 (4) | 5 (5) | 1 (1) | 2 (2) — includes initial, midcycle and terminal of any severity
Anger or irritability (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4) — any severity
oppositional (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1) | 4 (4) — any severity
mood lability (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) — any severity
# who withdrew due to AE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2) — any severity
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) — any severity
Agitation (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (4) — anyseverity

LIMITATIONS AND CAVEATS:
This was a very small study with a very heterogeneous sample. Further the two groups included very different proportions of intellectually disabled non-verbal participants which may influence assessment of benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No